CLINICAL TRIAL: NCT01899599
Title: A Double-blind, Placebo-controlled, Randomized, Phase 2 Study to Evaluate the Efficacy and Safety of Maintenance Therapy With PankoMab-GEX™ After Chemotherapy in Patients With Recurrent Epithelial Ovarian Carcinoma
Brief Title: PankoMab-GEX™ Versus Placebo as Maintenance Therapy in Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEXMab25201; 2013-000931-28 (EudraCT Number)
Record Dates: First submitted 2013-07-04; First posted 2013-07-15 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Epithelial Cancer Recurrent; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Ovarian Cancer; Maintenance Therapy
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — PankoMab-GEX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PankoMab-GEX (Experimental): 1700mg, i.v., q3w
  Interventions: Drug: PankoMab-GEX
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PankoMab-GEX — start dose 500mg at C0D1, maintenance dose 1700mg at CxD1, Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Gatipotuzumab
  Arms: PankoMab-GEX
Drug: Placebo — start dose matching 500mg at C0D1, maintenance dose matching 1700mg at CxD1, Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Placebo

SUMMARY:
Efficacy of PankoMab-GEX vs Placebo in maintaining a response to chemotherapy in advanced ovarian, fallopian tube or primary peritoneal cancer.

DETAILED DESCRIPTION:
The study is to evaluate the efficacy of PankoMab-GEX vs Placebo in maintaining response after 2nd to 5th line of chemotherapy in patients with epithelial ovarian or fallopian tube or primary peritoneal cancer. Patients must have responded to platinum based chemotherapy in a previous line, while the response to the most recent Pt-based chemotherapy must not have lasted more than 12 months. In addition the response between most recent 2 lines of chemotherapy prior start of study medication must not have lasted more than 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥18 years of age
2. Histologically-confirmed, TA-MUC1-positive, recurrent epithelial ovarian, or fallopian-tube cancer or primary peritoneal cancer with high-grade (Grade 2 or 3) serous features or a serous component
3. Availability of tumor tissue samples (slices or block) for immune-histological confirmation of TA-MUC1 status (tissue samples could also be stored for other further specified biomarker assessments)
4. Patients were to have received at least 2 lines but not more than 5 lines of chemotherapy prior to start of maintenance treatment; neo-adjuvant lines did not count as previous lines of treatment
5. Patients had to have a documented response to or SD following the most recent line of chemotherapy (any regimen and duration in accordance with local or international guidelines or within IEC-approved studies) and received the last dose of said chemotherapy ≤6 weeks prior to randomization (response to prior chemotherapy was defined as a PR/CR according to radiological response criteria and/or a confirmed decline in tumor marker CA125 ≥50% from the pre-treatment value for patients who had a pre-treatment value ≥2 x the upper limit of normal [ULN]; SD was defined as stable disease according to radiological response criteria with a confirmed lack of increase in tumor marker CA125 from the pre-treatment value for patients who had a pre-treatment value ≥2 × ULN and no clinical progression). Prior to randomization, CA125 had to be below the ULN, or CA125 levels were not to increase >15% within a time frame >7 days if above the ULN
6. Progression-free interval of ≤12 months immediately preceding the chemotherapy to which the patient had just responded
7. Sensitive or resistant to the most recent platinum-based chemotherapy preceding the chemotherapy to which the patient had just responded (sensitivity was thereby defined as a recurrence of disease >6 to ≤12 months after the end of platinum-based chemotherapy, and resistantance was defined as a recurrence of disease ≤6 months after the end of the platinum-based chemotherapy)
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
9. Recovered from all chemotherapy-related toxicities to Grade 1 or Grade 0 according to the NCI-CTCAE Version 4.0, with the exception of alopecia (any grade) and peripheral neuropathy (≤Grade 2)
10. Adequate bone marrow and hepatic function at Screening:

    * Hemoglobin ≥9 g/dL
    * White blood cell count ≥3.0 × 109/L
    * Absolute neutrophil count ≥1.5 × 109/L- Platelet count ≥100 × 109/L
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 × ULN (<5 × ULN in case of liver metastases)
    * Bilirubin <1.5 × ULN (<3 × ULN in case of liver metastases)
    * Creatinine <1.5 × ULN
11. Any patient with childbearing potential (i.e. not surgically sterile or post-menopausal for >1 year) had to use highly effective contraceptives with a Pearl index <1% according to the "Note for guidance on non-clinical safety studies for the conduct of human clinical trials and marketing authorization for pharmaceuticals" (CPMP/ICH/286/95) of the European Medicines Agency (EMA). (Although pregnancy was unlikely to occur in this patient population, any patient with childbearing potential had to be withdrawn from the study in the event of pregnancy)
12. Life expectancy >3 months
13. Ability and willingness to give written informed consent

Exclusion criteria:

1. Refractory to platinum-based chemotherapy (defined as remained progressive or became progressive under any previous platinum-based regimen)
2. Progression-free interval of >12 months after the most recent antecedent platinum-based chemotherapy regimen
3. Concomitant anti-tumor therapy or immunotherapy
4. Treatment with monoclonal antibodies or investigational agents ≤30 days before randomization (prior anti-MUC1 therapy was not permitted at any time)
5. Limited-field radiotherapy ≤30 days before randomization (extensive prior radiotherapy during or following the last line of chemotherapy was not permitted; radiotherapy prior to the last line of chemotherapy was permitted)
6. Prior allergic reaction to a monoclonal antibody, Grade 3 IRR or any Grade 4 reaction to a monoclonal antibody
7. Known sensitivity to any component of the test product
8. Contraindication to the pre-medication used in this study (paracetamol/acetaminophen, H1 and/or H2 receptor antagonists, or steroids)
9. Clinical evidence of brain metastasis or leptomeningeal involvement
10. Patients with second primary cancer, except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, ductal carcinoma in situ, Stage 1 Grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years
11. Primary or secondary immune deficiency
12. Clinically active infections >Grade 2 using NCI-CTCAE version 4.0
13. Active hepatitis B or C or infection with human immunodeficiency virus (HIV)
14. Myocardial infarction within 6 months prior to Screening
15. Symptomatic congestive heart failure (New York Heart Association Grade 3 or 4), unstable angina pectoris within 6 months prior to Screening, significant cardiac arrhythmia or history of stroke or transient ischemic attack within 1 year prior to Screening
16. Prior or planned major surgery within 30 days prior to randomization and/or incomplete recovery from prior surgery
17. Concomitant use of systemic steroids, except for inhaled, topical or nasal application within 30 days prior to randomization (steroids used for pre-medication were permitted)
18. Active drug or alcohol abuse
19. Any uncontrolled medical condition that could have put the patient at high risk during treatment with an investigational drug, including unstable diabetes mellitus, vena cava syndrome, or chronic symptomatic respiratory disease
20. Pregnancy or lactation
21. Legal incompetence, limited legal competence, or detainment in an institution for official or legal reasons
22. Receipt of any other investigational medicinal product within the last 30 days before randomization or any previous PankoMab-GEX™ administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Progression free survival | from baseline till progression of disease or death
  PFS will be determined by radiographic progression based on modified RECIST 1.1 or death of any cause.

SECONDARY OUTCOMES:
To assess the safety and tolerability of maintenance therapy with single-agent PankoMab-GEX™ compared to placebo in patients with metastatic or recurrent ovarian or fallopian tube carcinoma or primary peritoneal carcinoma. | from randomization until end of treatment
  Safety will be determined on the occurrence of infusion-related reactions (IRR), treatment emergent adverse events (TEAE) and treatment emergent serious adverse events (TESAE).
Patient reported outcome | from randomization until end of treatment
  To evaluate the quality of life (QoL) and other health and health-economy related outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ledermann, MD, Principal Investigator — UCL Cancer Institute, 90 Tottenham Court Road, London W1T 4TJ, UK
Locations (37):
- Germany (5):
  - Investigator, Berlin
  - Investigator, Kiel
  - Investigator, Munich
  - Investigator, Regensburg
  - Investigator, Stuttgart
- Hungary (3):
  - Investigator, Budapest
  - Investigator, Debrecen
  - Investigator, Szeged
- Italy (3):
  - Investigator, Meldola
  - Investigator, Milan
  - Investigator, Rome
- Poland (6):
  - Investigator, Bydgoszcz
  - Investigator, Gdansk
  - Investigator, Lublin
  - Investigator, Olsztyn
  - Investigator, Poznan
  - Investigator, Rzeszów
- Romania (6):
  - Investigator, Brasov
  - Investigator, Bucharest
  - Investigator, Cluj-Napoca
  - Investigator, Craiova
  - Investigator, Oradea
  - Investigator, Timișoara
- Russia (8):
  - Investigator, Kazan'
  - Investigator, Moscow
  - Investigator, Oryol
  - Investigator, Pyatigorsk
  - Investigator, Rostov-on-Don
  - Investigator, Saint Petersburg
  - Investigator, Volgograd
  - Investigator, Yaroslavl
- Spain (3):
  - Investigator, Barcelona
  - Investigator, Madrid
  - Investigator, Valencia
- United Kingdom (3):
  - Investigator, London
  - Investigator, Northwood
  - Investigator, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ledermann JA, Zurawski B, Raspagliesi F, De Giorgi U, Arranz Arija J, Romeo Marin M, Lisyanskaya A, Poka RL, Markowska J, Cebotaru C, Casado Herraez A, Colombo N, Kutarska E, Hall M, Jacobs A, Ahrens-Fath I, Baumeister H, Zurlo A, Sehouli J. Maintenance therapy of patients with recurrent epithelial ovarian carcinoma with the anti-tumor-associated-mucin-1 antibody gatipotuzumab: results from a double-blind, placebo-controlled, randomized, phase II study. ESMO Open. 2022 Feb;7(1):100311. doi: 10.1016/j.esmoop.2021.100311. Epub 2021 Dec 15. PMID 34920291